CLINICAL TRIAL: NCT06513338
Title: A Single Center, Open-label, Single Arm Phase II Trial of the Efficacy and Safety of Complement C5 Monoclonal Antibody in the Treatment of Anti-glomerular Basement Membrane Disease
Brief Title: Complement C5 mAb in the Treatment of Anti-GBM Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Zhao CUI, Dr., Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C5mAb in anti-GBM disease
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Autoimmune Diseases
Keywords: complement C5; crescentic glomerulonephritis; anti-GBM disease; complement inhibition
MeSH Terms: conditions — Autoimmune Diseases; Anti-Glomerular Basement Membrane Disease | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eculizumab (Experimental): C5 monoclonal treatment plus standard treatment
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — eculizumab 900mg iv. per week for 4 weeks, then 1200mg every two weeks for 8 weeks

SUMMARY:
Anti-GBM disease is the most severe form of glomerulonephritis. Despite of the standard treatment including plasmapheresis and immunosuppressant, 70% of the patients still go into end-stage kidney disease. Complement has been shown to participate in the pathogenesis of anti-GBM disease. This study aims to the investigate the therapeutic effects and safety of C5 monoclonal antibody in the treatment of anti-GBM disease.

DETAILED DESCRIPTION:
Anti-glomerular basement membrane (anti-GBM) disease is the most severe form of autoimmune glomerulonephritis, characterized by the production of autoantibodies targeting the components of basement membrane within the kidney and/or the lung.Patients with anti-GBM disease typically present rapidly progressive glomerulonephritis, and often accompanied by lung hemorrhage. The hallmark of the disease is the linear deposition of IgG along the GBM on kidney biopsy. Complement activation is a pivotal step for kidney injuries during the development of human anti-GBM disease. Our previous study showed that the The levels of plasma SC5b-9 and urinary C5a were positively correlated with the serum creatinine at presentation and the percentage of crescents in glomeruli. Eculizumab is a recombinant humanized monoclonal antibody that specifically binds to a C5 terminal complement and inhibits the cleavage of C5 to C5a and C5b through complement activation. There are a few case reports showing therapeutic effects in anti-GBM disease. This trial will aim to evaluate the efficacy and safety of Eculizumab plus standard treatment in anti-GBM disease.

ELIGIBILITY:
Inclusion Criteria

1. Positive circulating anti-GBM antibody, with proteinuria or hematuria or any clinical signs of kidney injuries.
2. And or kidney biopsy showed typical IgG linear deposition along the GBM
3. At least 18 years old

Exclusion Criteria

1. Allergic to eculizumab, mouse protein or the investigational drug and any of its excipients;
2. Uncontrolled meningococcal infection,or those who have not received meningitis prophylactic antibiotic treatment or meningitis vaccination;
3. Diagnosis of anti-GBM disease for more than 12 weeks before signing the informed consent form;
4. Pregnant or lactating
5. Received investigational drug within 30 days or 4 half-lives (whichever is longer) prior to screening;
6. Other serious poorly controlled comorbid diseases that affect the compliance of the trial protocol or the interpretation of results within 3 months prior to screening, including cardiovascular and cerebrovascular diseases, lung disease, etc.;
7. Presence of any medical history or disease that, in the opinion of the investigator, may expose the patient's participation in the study to an unacceptable risk;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
kidney prognosis | 6 months after the first infusion of eculizumab
  ESKD (dialysis dependent) or kidney translation

SECONDARY OUTCOMES:
Changes in glomerular filtration rate (eGFR); | from baseline to study completion, an average of 1 year
  Change in level of estimated Glomerular Filtration Rate (eGFR) as measured by laboratory testing, reported in mL/min/1.73m².
Changes in serum creatinine | from baseline to study completion, an average of 1 year
  Change in concentration of serum creatinine as measured by laboratory testing, reported in µmol/L
Changes in blood urine nitrogen (BUN) | from baseline to study completion, an average of 1 year
  Change in concentration of Blood Urea Nitrogen (BUN) as measured by laboratory testing, reported in mmol/L
side effects of eculizumab | at 6 months
  The number of participants experiencing any adverse events determined by the investigator to be related to eculizumab treatment.

OTHER OUTCOMES:
kidney function recovery | 6 months after the first eculizumab infusion
  Kidney recovery was defined as independence from kidney replacement therapy (KRT, such as dialysis) lasting at least 12 weeks during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Cui, Principal Investigator — PKUFH
Locations (1):
- Peking University First Hospital, Beijing, China